CLINICAL TRIAL: NCT06388408
Title: Effects of Sufentanil Delivered With Target Controlled Infusion (TCI) on Patient State Index Values, Electroencephalographic Spectrum and Analgesia Nociception Index During Total Intravenous Anesthesia With Propofol TCI
Brief Title: Effects of Sufentanil Target Controlled Infusion on Patient State Index Values and Electroencephalographic Spectrum During Total Intravenous Anesthesia With Propofol
Status: Completed | Type: Observational
Sponsor: University of Padova (Other)
Responsible Party: Principal Investigator, Federico Linassi, MD, prinicpal investigator, University of Padova
Other Study IDs: SufMAST
Record Dates: First submitted 2024-03-24; First posted 2024-04-29 (Actual); Last update posted 2024-10-24 (Actual); Status verified 2024-10

CONDITIONS: Anesthesia Brain Monitor; Sufentanil; Target Controlled Infusion

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Sufentanil Target Controlled infusion (TCI, Gepts model) effects on Neuromonitoring during Total Intravenous Anesthesia (TIVA) with Propofol TCI (Eleveld model) has not been investigate yet.

Authors aim to investigate its effect on Patient State index (PSi), the power spectrum EEG, the Analgesia Nociception Index (ANI) nad pupillometry values during maintenance durin TIVA-TCI with Propofol and Sufentanil.

DETAILED DESCRIPTION:
Sufentanil Target Controlled infusion (TCI, Gepts model) effects on Neuromonitoring during Total Intravenous Anesthesia (TIVA) with Propofol TCI (Eleveld model) has not been investigate yet.

Authors aim to investigate its effect on Patient State index (PSi), the power spectrum EEG, the Analgesia Nociception Index (ANI) and pupillometry values during maintenance during TIVA-TCI with Propofol and Sufentanil.

ELIGIBILITY:
Inclusion Criteria:

* Undergo general anaesthesia with Targeted Controlled Infusion of Propofol (Eleveld model) and Sufentanil (Gepts model)

Exclusion Criteria:

* Neurological disease
* Psychiatric disease
* Obesity
* Regional anesthesia performed

Ages: 18 Years to 90 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Women undergoing brast cancer surgery with general anesthesia with Propofol and SufentanilTCI will be recruited
Sampling Method: Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2024-05-05 (Actual); Primary Completion 2024-09-15 (Actual); Study Completion 2024-09-30 (Actual)

PRIMARY OUTCOMES:
Effects of Sufentanil on Patient State index (PSi) during stable Propofol general anesthesia | PSi values and Sufentanil Target Controlled Infusion (TCI) concentrations will be monitored during all the time of surgery
  Evaluate if sufentanil variations during general anesthesia has an impact on the PSi values
Effects of Sufentanil on Electroencephalogram (EEG) power spectrum during stable Propofol general anesthesia | EEG power spectrum and Sufentanil Target Controlled Infusion (TCI) concentrations will be monitored during all the time of surgery
  Evaluate if sufentanil variations during general anesthesia has an impact on the EEG power spectrum
Effects of Sufentanil on Analgesia Nociception Index (ANI) during stable Propofol general anesthesia | ANI values and Sufentanil Target Controlled Infusion (TCI) concentrations will be monitored during all the time of surgery
  Evaluate if sufentanil variations during general anesthesia has an impact on the ANI values

SECONDARY OUTCOMES:
Analgesia Nociception Index (ANI) values and postoperative pain | Numeric Rating Scale (NRS) will be evaluated after the end of surgery and 24 hours after the end of surgery and compared to ANI values after 24 hours
  Evaluate if different ANI values at the same Sufentanil concentrations has an impact on postoperative pain
Patient State Index (PSi) values and postoperative delirium | Confusion assessment method (CAM) test for delirium will be performed after the end of surgery and compared to PSi values after 24 hours
  Evaluate if different PSi values at the same Sufentanil concentrations has an impact on postoperative pain
Analgesia Nociception Index (ANi) values and postoperative nausea and vomiting | Nausea and vomiting occurrence will be detected hours atend of surgery and compared to ANI values after 24 hours
  Evaluate if different ANi values at the same Sufentanil concentrations has an impact on postoperative nausea and vomiting.

CONTACTS AND LOCATIONS:
Overall Officials: Federico Linassi, MD, Principal Investigator — University of Padova
Locations (1):
- Treviso Regional Hospital, Treviso, TV, Italy

IPD SHARING:
Plan to Share IPD: Undecided